CLINICAL TRIAL: NCT02003027
Title: Endomyocardial Botulinum Toxin Injection Can Decrease the Number of Episodes of VT Storm: Pilot Study
Brief Title: Botulinum Toxin Injection to Prevent VT Storm
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT_VT Storm
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: VT Storm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BT injection (Experimental)
  Interventions: Drug: BT injection

INTERVENTIONS:
Drug: BT injection

SUMMARY:
The aim of this prospective non-randomized study was to assess the efficacy and safety of endomyocardial botulinum toxin injection in left ventricle for preventing episodes of VT Storm.

ELIGIBILITY:
Inclusion Criteria:

* 3 or more episodes of ventricular tachycardia within 24 hours

Exclusion Criteria:

* Failure to provide informed consent.
* Non-cardiac illness with a life expectancy of less than 3 year
* Non-cardiac illness imposing substantial operative mortality
* Current participation in another clinical trial in which a patient is taking an investigational drug or receiving an investigational medical device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
number of episodes of VT Storm | 1 year

SECONDARY OUTCOMES:
serious adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru